CLINICAL TRIAL: NCT06855771
Title: A Multicenter, Randomized, Open-label, Phase 2 Study Evaluating the Safety and Efficacy of BMS-986504 Monotherapy in Participants With Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) With Homozygous MTAP Deletion After Progression on Prior Therapies
Brief Title: A Study of BMS-986504 in Participants With Pre-treated Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) With Homozygous MTAP Deletion (MountainTAP-9)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA240-0009; 2024-519814-29 (Other: EU CTR); U1111-1315-9473 (Other: WHO)
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: BMS-986504 Dose 1 (Experimental)
  Interventions: Drug: BMS-986504
- Arm B: BMS-986504 Dose 2 (Experimental)
  Interventions: Drug: BMS-986504

INTERVENTIONS:
Drug: BMS-986504 — Specified dose on specified days
  Other Names: MRTX1719

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BMS-986504 monotherapy in participants with advanced or metastatic Non-small Cell Lung Cancer (NSCLC) with homozygous MTAP deletion after progression on prior therapies.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed diagnosis of NSCLC and homozygous MTAP deletion detected in tumor tissue and willingness to provide archival/fresh samples at screening for central MTAP status confirmation.
* Advanced or metastatic NSCLC not amenable to curative therapies after progression on prior therapies at the time of enrollment (based on the American Joint Committee on Cancer, Ninth Edition).
* At least 1 measurable lesion as per RECIST v1.1.
* Documented radiographic disease progression on or after the most recent line of treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Participant must be ≥ 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place) at the time of signing the ICF.
* Capability to swallow tablets intact (without chewing or crushing).

Exclusion Criteria

* Active brain metastases or carcinomatous meningitis.
* History of gastrointestinal disease or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications.
* Prior treatment with a PRMT5 or MAT2A inhibitor.
* Known severe hypersensitivity to study treatment and/or any of its excipients.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve Objective Response (OR) utilizing the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 3 years after the last participant's last dose of study treatment
  OR is defined as confirmed complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Number of participants who achieve disease control (DC) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
  DC is defined as Best Overall Response (BOR) of confirmed CR, confirmed PR, or stable disease (SD)
Number of participants who achieve clinical benefit (CB) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
  CB is defined as BOR of confirmed CR, confirmed PR, or SD for at least 6 months after start of treatment
Duration of response (DOR) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
  DOR is defined as the time between the date of the first documentation of objective tumor response (CR or PR) and the date of disease progression or to death from any cause (whichever occurs first)
Progression-free survival (PFS) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
  PFS is defined as the time between randomization and the date of disease progression or death from any cause (whichever occurs first)
Time to objective response (TTOR) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
  TTOR is defined as the time between randomization to the date of the first documentation of objective tumor response (CR or PR)
Number of participants with adverse events (AE) | Up to 28 days after the last dose of study treatment
Number of participants with Serious AEs (SAEs) | Up to 28 days after the last dose of study treatment
Number of participants with AEs leading to dose interruption, reduction, or discontinuation | Up to 28 days after the last dose of study treatment
Number of deaths | Up to 28 days after the last dose of study treatment
Number of participants who achieve Objective Response (OR) as assessed by RECIST v1.1 | Up to 3 years after the last participant's last dose of study treatment
Overall Survival (OS) | Up to 3 years after the last participant's last dose of study treatment
  OS is defined as the time between the randomization/the start of treatment to death due to any cause
Change from baseline in cancer-related symptoms and health-related quality of life as assessed by the Non-small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) total score and symptom score | Up to 28 days after the last dose of study treatment
Change from baseline in cancer-related symptoms and health-related quality of life as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core Function Global Health Status functional scale score | Up to 28 days after the last dose of study treatment
Change from baseline in cancer-related symptoms and health-related quality of life as assessed by the EORTC-QLQ-F17 quality-of-life (QoL) functional scale score | Up to 28 days after the last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (71):
- United States (12):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Local Institution - 0099, Boise, Idaho
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0079, Shirley, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutchison Cancer Center, Seattle, Washington
  - Local Institution - 0084, Milwaukee, Wisconsin
- Australia (4):
  - GenesisCare - Campbelltown, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - GenesisCare - St Andrew's, Adelaide, South Australia
- China (9):
  - Local Institution - 0039, Beijing, Beijing Municipality
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Local Institution - 0056, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Local Institution - 0044, Linyi, Shandong
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
- France (9):
  - Local Institution - 0045, Marseille, Bouches-du-Rhône
  - Chu Grenoble Alpes, La Tronche, Isère
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron, Rhône
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Local Institution - 0107, Paris
  - Hôpital Tenon, Paris
  - Groupe hospitalier Paris saint Joseph, Paris, Île-de-France Region
- Germany (5):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main, Hesse
  - Krankenhaus Martha-Maria Halle-Dölau, Halle, Saxony-Anhalt
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (7):
  - AOU della Campania Luigi Vanvitelli, Napoli, Campania
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
- Japan (3):
  - Local Institution - 0092, Kashiwa, Chiba
  - Local Institution - 0094, Sendai, Miyagi
  - Local Institution - 0093, Hirakata, Osaka
- Poland (2):
  - Mazowiecki Szpital Onkologiczny, Wieliszew, Masovian Voivodeship
  - Local Institution - 0064, Prabuty
- Romania (7):
  - Institutul Oncologic Bucuresti "Prof. Dr. Alexandru Trestioreanu", Bucharest, București
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Local Institution - 0040, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - S.C. Centrul de Oncologie Euroclinic S.R.L., Iași
  - Institutul Regional de Oncologie, Iași
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, Hospitalet, Barcelona [Barcelona]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna, Solna, Stockholms Län [se-01]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands Län [se-14]
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Sarah Cannon Research Institute UK, London, London, City of
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06855771.html